CLINICAL TRIAL: NCT03883399
Title: Awareness of Practice and Comparison With Best Evidence in Surgical Site Infection Prevention in Colorectal Surgery
Brief Title: Survey on Practice and Comparison With Best Evidence in Surgical Site Infection Prevention in Colorectal Surgery
Acronym: PREVISQCOR
Status: Completed | Type: Observational
Sponsor: Hospital de Granollers (Other)
Responsible Party: Principal Investigator, Josep Maria Badia, Prof, Hospital de Granollers
Other Study IDs: PREVISQCOR-19
Record Dates: First submitted 2019-03-11; First posted 2019-03-20 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Surgery; Surgical Site Infection
Keywords: Surgical Site Infection; Prevention; Survey; Colorectal surgery; Guidelines
MeSH Terms: conditions — Surgical Wound Infection | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal surgeons: Survey among Spanish colorectal surgeons
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey among colorectal surgeons

SUMMARY:
Web-based survey to colorectal surgeons assessing knowledge, beliefs and practices regarding the use of preventative measures for SSI.

DETAILED DESCRIPTION:
A web-based survey (SurveyMonkey©; https://es.surveymonkey.com/r/FBVR59C) to the members of the Colorectal Chapter of the Spanish Association of Surgeons (AEC) and the Spanish Association of Coloproctology (AECP). A link to the web page containing the survey is disseminated via email, newsletter and Twitter.

A board from the Surgical Infection Section did a review of evidence and previous guidelines to be used in the evaluation of the results. The most recent clinical practice guidelines have been analysed. Furthermore, an extensive review of specific measures for colorectal surgery has been published and used for evaluation. According to the review, the preventive measures analysed in the survey have been distributed into two groups: high or low level of evidence.

The survey aim to assess knowledge, beliefs, and practices of attending colorectal surgeons on preventative measures including mechanical bowel preparation (MBP), oral antibiotic prophylaxis and the use of drains. Furthermore, the questions address the level of accordance between their beliefs and the protocols or the usual practice of their units. The agreement rate between the beliefs and usual practice of all respondents will be calculated on a scale from 0 to 100. For discussion, the responses on the implementation of major surgical site infection (SSI) prevention measures will be compared with the recommendations of the expert group. Other questions are related to the types of complications that surgeons believe are prevented by the use of oral antibiotic prophylaxis or MBP, reasons for not using either of them, type of oral and systemic antibiotics and cathartics used, and strategies already in place or that should be implemented to reduce SSI rates at respondents' hospitals.

The results will be expressed in percentages on the total answers obtained. Responses will be entered into a computerized database that will be analysed using the SPSS program (v.10.0, Chicago, IL, USA). The results will be analysed using the chi-square test with statistical significance defined as p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal surgeons members of the Colorectal Chapter of the Spanish Association of Surgeons (AEC) and the Spanish Association of Coloproctology (AECP)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Members of the Colorectal Chapter of the Spanish Association of Surgeons (AEC) and the Spanish Association of Coloproctology (AECP)
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Awareness of practice - Percentage of responders who use each preventive measures for surgical site infection | 2019
  Percentage of responders who use each preventive measures for surgical site infection (including mechanical bowel preparation and oral antibiotic prophylaxis), compared to their beliefs and knowledge of scientific evidence.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Badia, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Fundació Privada Hospital Asil de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided